CLINICAL TRIAL: NCT04569747
Title: 20-347 NCT Number Title A Single Arm Phase II Study of ADjuvant Endocrine Therapy, Pertuzumab, and Trastuzumab for Patients With Anatomic Stage I Hormone Receptor-positive, HER2-positive Breast Cancer (ADEPT)
Brief Title: A Single Arm Phase II Study of ADjuvant Endocrine Therapy, Pertuzumab, and Trastuzumab for Patients With Anatomic Stage I Hormone Receptor-positive, HER2-positive Breast Cancer
Acronym: ADEPT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Adrienne G. Waks, Sponsor Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-347
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: HER2-positive Breast Cancer; Invasive Carcinoma of the Breast; Breast Cancer; Node Negative Breast Cancer; Micrometastasis Breast Cancer; Hormone Receptor Positive Breast Cancer
Keywords: HER2-positive Breast Cancer; Invasive Carcinoma of the Breast; Breast Cancer; Node Negative Breast Cancer; Micrometastasis Breast Cancer; Hormone Receptor Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Anastrozole; exemestane; Tamoxifen; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PERTUZUMAB + TRASTUZUMAB + ADJUVANT ENDOCRINE THERAPY (Experimental): Study treatment will be administered in 21-day (3- week, +/- 3 days) cycles for one year (18 cycles).
  * Trastuzumab + Pertuzumab SC fixed dose combination
  * Hormonal therapy- oral, daily per cycle (may add LHRH agonist per investigator discretion)
  Interventions: Combination Product: Pertuzumab+TRASTUZUMAB; Drug: ADJUVANT ENDOCRINE THERAPY

INTERVENTIONS:
Combination Product: Pertuzumab+TRASTUZUMAB — Trastuzumab + pertuzumab SC FDC (PHESGO) will be administered on Day 1 of each 21-day cycle , subcutaneous, fixed dose
  Other Names: PHESGO
Drug: ADJUVANT ENDOCRINE THERAPY — Oral, daily per cycle
  Other Names: Letrozole; Anastrozole; Exemestane; Tamoxifen; Leuprolide, or other LHRH agonist (per investigator discretion)

SUMMARY:
This research study is studying a combination of HER2-directed therapies (trastuzumab and pertuzumab) and hormonal therapy as a treatment after surgery for hormone receptor positive breast cancer.

The study drugs involved in this study are:

* A combination of trastuzumab and pertuzumab given as an injection under the skin (PHESGO)
* Hormonal (endocrine) Treatment

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility and study treatment including laboratory evaluations, physical exams, questionnaires, and follow up visits.

* Participants will receive HER2-directed treatment for 1 year and hormonal therapy for approximately 5 years.
* It is expected that about 375 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug combination to learn whether the drug works in treating a specific disease. "Investigational" means that the drug combination is being studied.

The drugs trastuzumab and pertuzumab are both monoclonal antibodies, which are disease-fighting proteins made by cloned immune cells. The U.S. Food and Drug Administration (FDA) has approved trastuzumab, pertuzumab, and trastuzumab + pertuzumab subcutaneous fixed dose combination (PHESGO) as treatment for HER2 positive breast cancer. The FDA has also approved hormonal therapies as treatment for hormone receptor positive breast cancer.

.

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive T1 histologically confirmed invasive carcinoma of the breast. Patients must have node-negative (N0) or micrometastases (N1mi) breast cancer according to the AJCC 8th edition anatomic staging table.

  * If the patient has had a negative sentinel node biopsy, then no further axillary dissection is required, and the patient is determined to be node-negative. Axillary nodes with single cells or tumor clusters ≤ 0.2 mm by either H&E or immunohistochemistry (IHC) will be considered node-negative.
  * Any axillary lymph node with tumor clusters between 0.02 and 0.2cm is considered a micrometastasis. Patients with a micrometastasis are eligible. An axillary dissection is not required to be performed in patients with a micrometastasis found by sentinel node evaluation. In cases where the specific pathologic size of lymph node involvement is subject to interpretation, the Sponsor-Investigator will make the final determination as to eligibility. The investigator must document approval in the patient medical record.
  * Patients who have one or more foci of T1aN0, ER+ (defined as >10%), HER2-negative cancer in the ipsilateral breast, in addition to their primary HER2-positive tumor, are eligible.
* For unifocal disease, all invasive disease must have been tested for ER and PR (for multifocal disease, see below). Either ER or PR must be positive, defined as ER ≥10% or PR ≥10%. ER- and PR-assays should be performed by immunohistochemical methods according to the local institution standard protocol.
* HER2-positive by ASCO CAP 2018 guidelines.
* Bilateral breast cancers that individually meet eligibility criteria are allowed.
* Patients with multifocal or multicentric disease are eligible as long as each tumor individually meets eligibility criteria.
* Patients with a history of ipsilateral DCIS are eligible as long as the patient has not received prior hormonal therapy. Patients with a history of contralateral DCIS are not eligible unless contralateral DCIS was diagnosed at least 15 years ago
* ≤ 95 days between the date of protocol registration and the patient's most recent breast surgery for this breast cancer
* Patients must have undergone definitive breast surgery for the current malignancy. All tumor should be removed by either a modified radical mastectomy or a segmental mastectomy (lumpectomy), with either a sentinel node biopsy or axillary dissection

  -- All margins should be clear of invasive cancer or DCIS (i.e. no tumor on ink). The local pathologist must document negative margins of resection in the pathology report. If all other margins are clear, a positive posterior (deep) margin is permitted, provided the surgeon documents that the excision was performed down to the pectoral fascia and all tumor has been removed. Likewise, if all other margins are clear, a positive anterior (superficial; abutting skin) margin is permitted provided the surgeon documents that all tumor has been removed. Radiation therapy to the conserved breast is required.
* Patients may have received up to 8 weeks of hormonal therapy as adjuvant treatment for this cancer. Patients should otherwise not have received prior hormonal therapy with the exception that hormonal therapy administered for less than 8-week duration at least 15 years ago is allowed.
* Prior oophorectomy (including for cancer therapy) is allowed.
* Patients undergoing breast conservation therapy (i.e. lumpectomy) must not have any contraindications to radiation therapy.
* Patients who have participated in a window study (treatment with an investigational agent prior to surgery for ≤2 weeks) are eligible. Patients must have discontinued the investigational agent at least 14 days before participation in this study.
* Men and women with any menopausal status ≥18 years of age
* ECOG Performance Status 0 or 1
* Participants must have normal organ and marrow function as defined below:

  * ANC ≥ 1000/mm3
  * hemoglobin ≥8 g/dl
  * platelets ≥ 75,000/mm3
  * AST and ALT both <5x institutional ULN
  * Total bilirubin ≤ 1.5 mg/dL. For patients with Gilbert syndrome, the direct bilirubin should be <institutional ULN
  * Serum creatinine ≤ 2.0 mg/dL OR calculated GFR ≥ 30mL/min
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Post-menopausal patients must meet one of the following criteria:

  * Prior bilateral ovariectomy/oophorectomy
  * Age ≥ 60 years
  * Age < 60 years with intact uterus and amenorrhoeic for ≥ 12 consecutive months prior to chemotherapy and/or endocrine therapy exposure (medication-induced amenorrhea is not acceptable to meet this criterion)
  * Age < 60 years hysterectomized and FSH and plasma estradiol levels in the postmenopausal range according to local policies prior to chemotherapy and/or endocrine therapy exposure.
* Willingness to discontinue contraceptive hormonal therapy, e.g. birth control pills, prior to registration and while on study
* Premenopausal patients with intact uterus must have a negative serum or urine pregnancy test, including women who have had a tubal ligation and women less than 12 months from their last menstrual period.
* Women of childbearing potential and men with partners of childbearing potential must be willing to use one highly effective form of nonhormonal contraception or two effective forms of nonhormonal contraception by the patient and/or partner and continue its use for the duration of the study treatment and for 7 months after the last dose of antibody treatment and 3 months after the last dose of hormonal treatment.
* Patients must be willing and able to sign informed consent.
* Patients must be willing to provide archival tissue for research purposes.
* If patient is English-speaking, must be willing to fill out patient questionnaires.

Exclusion Criteria:

* Neoadjuvant or adjuvant chemotherapy for this breast cancer prior to enrollment is prohibited.
* Any of the following due to teratogenic potential of the study drugs:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragms, IUDS, surgical sterilization, abstinence, etc). Hormonal birth control methods are not permitted.
  * Men who are unwilling to employ adequate contraception (condoms, surgical sterilization, abstinence, etc).
* Participants who are receiving any other investigational agents for treatment of breast cancer, unless specific approval is obtained from the Sponsor-Investigator.
* Locally advanced tumors at diagnosis, including tumors fixed to the chest wall, peau d'orange, skin ulcerations/nodules, or clinical inflammatory changes (diffuse brawny cutaneous induration with an erysipeloid edge)
* Patients with a history of previous invasive breast cancer.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances:

  * Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy.
  * individuals with the following cancer are eligible regardless of when they were diagnosed and treated: cervical cancer in situ, and non-melanoma cancer of the skin.
* Intercurrent illness including, but not limited to: ongoing or active, unresolved systemic infection, renal failure requiring dialysis, active cardiac disease, prior myocardial infarction (asymptomatic changes on EKG suggestive of old MI is not an exclusion), history of CHF, current use of any therapy specifically for CHF, uncontrolled hypertension, significant psychiatric illness, or other conditions that in the opinion of the investigator limit compliance with study requirements.

Time and Motion Substudy Eligibility:

* Participant must be enrolled at Dana-Farber Cancer Institute
* Participant must not have discontinued pertuzumab following treatment cycle 1
* Participant must be able to tolerate subcutaneous administration following cycle 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease Free Survival at 3 Years | 3 Years
  Kaplan-Meier estimates of iDFS will be estimated and plotted with the corresponding 95% confidence intervals.
  from the time of randomization until the occurrence of the first of the following events: invasive local/regional recurrence, Contralateral invasive breast cancer, Distant recurrence, Death from any cause

SECONDARY OUTCOMES:
Invasive Disease Free Survival at 7 Years | 7 years
  Kaplan-Meier estimates of iDFS will be estimated and plotted with the corresponding 95% confidence intervals.
  from the time of randomization until the occurrence of the first of the following events: invasive local/regional recurrence, Contralateral invasive breast cancer, Distant recurrence, Death from any cause
Invasive Disease Free Survival at 10 Years | 10 years
  Kaplan-Meier estimates of iDFS will be estimated and plotted with the corresponding 95% confidence intervals.
  from the time of randomization until the occurrence of the first of the following events: invasive local/regional recurrence, Contralateral invasive breast cancer, Distant recurrence, Death from any cause
Recurrence-free interval (RFI) at 3 Years | 3 Years
  RFI will be estimated and plotted with the corresponding 95% confidence intervals, using Kaplan-Meier estimates for the study as a whole and for subgroups of patients determined by intrinsic subtype (HER2-enriched, luminal, basal Time of randomization until the occurrence of the first of the following events:Invasive local/regional recurrence, Distant recurrence, Death from breast cancer
Recurrence-free interval (RFI) at 7 Years | 7 Years
  RFI will be estimated and plotted with the corresponding 95% confidence intervals, using Kaplan-Meier estimates for the study as a whole and for subgroups of patients determined by intrinsic subtype (HER2-enriched, luminal, basal Time of randomization until the occurrence of the first of the following events:Invasive local/regional recurrence, Distant recurrence, Death from breast cancer
Recurrence-free interval (RFI) at 10 Years | 10 Years
  RFI will be estimated and plotted with the corresponding 95% confidence intervals, using Kaplan-Meier estimates for the study as a whole and for subgroups of patients determined by intrinsic subtype (HER2-enriched, luminal, basal Time of randomization until the occurrence of the first of the following events:Invasive local/regional recurrence, Distant recurrence, Death from breast cancer
Breast cancer-specific survival (BCSS) at 3 Years | 3 Years
  defined as the time period between randomization and death due to breast cancer.
Breast cancer-specific survival (BCSS) at 7 Years | 7 Years
  defined as the time period between randomization and death due to breast cancer.
Breast cancer-specific survival (BCSS) at 10 Years | 10 Years
  defined as the time period between randomization and death due to breast cancer.
Overall survival | randomization and death. Surviving patients classified as lost-to-follow-up or having withdrawn consent to be followed will be censored at their date of last contact or withdrawal of consent to be followed, whichever occurs first up to 10 years
  OS will be estimated and plotted with the corresponding 95% confidence intervals, using Kaplan-Meier estimates for the study as a whole and for subgroups of patients determined by intrinsic subtype (HER2-enriched, luminal, basal).
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | baseline to 5 Years
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting
Total patient chair time of drug administration | baseline to 18 Months
  Mean difference will be estimated between HP FDC SC and IV admin of HP in sub-study

OTHER OUTCOMES:
Patient-reported hormonal therapy adherence | 5 years
  assessed by Voils questionnaire. Responses to survey items will be summarized using means or proportions depending on the nature of the questions.
FACT B | baseline to 18 Months
  The FACT-B includes the FACT-G, a 27-item generic cancer questionnaire and a 10- item breast cancer specific module. Responses to survey items will be summarized by means or proportions depending on the nature of the items
Rotterdam symptom checklist, | baseline to 18 Months
  The Activity Level Scale Domain from the RSCL is an 8-item scale designed to measure whether the respondent can perform a series of activities at the present time. Items are summed to produce an overall score, with higher scores representing better functioning.
  Responses to survey items will be summarized by means or proportions
WPAI-SHP-Work Productivity | baseline to 18 Months
  The WPAI was created as a patient-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to general health (WPAI:GH) or a specific health problem (WPAI:SHP). The 6 questions in the WPAI questionnaire were generated from three main sources Responses to survey items will be summarized by means or proportions depending on the nature of the items
COST-Financial Toxicity | baseline to 18 Months
  There is increasing recognition of the profound importance of the financial strain on patients created by cancer diagnosis and therapies. The COST (Comprehensive Score for financial Toxicity) measure has been developed and validated as a mechanism to assess financial stress related to cancer diagnosis and treatment Responses to survey items will be summarized by means or proportions
Patient Acceptance of subcutaneous therapy (HPASQ-SC) | baseline to 18 Months
  The HPASQ-SC (Appendix C) is a tool to measure patient-reported outcomes regarding patient acceptance of subcutaneous therapy. It was developed and underwent validity testing in a cohort of patients receiving subcutaneous rituximab for lymphoma. The HPASQ-SC contains questions related to two main concepts (treatment satisfaction and impact of treatment administration) and eight sub-concepts: overall preference/satisfaction; convenience; confidence; bothersome-ness; physical impact; psychological impact; impact on activities of daily life; and impact on the interaction with healthcare providers.21
  Responses to survey items will be summarized by means or proportions
Patient treatment experience time | baseline to 18 Months
  Comparing FDC HP to IV HP in sub-study
Patient drug administration time | baseline to 18 Months
  Comparing FDC HP to IV HP in sub-study
Pharmacist time commitment for drug preparation | baseline to 18 Months
  Comparing FDC HP to IV HP in sub-study

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne C Waks, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (32):
- United States (32):
  - Stamford Hospital, Stamford, Connecticut
  - University of Miami- Sylvester Comprehensive Cancer Center, Miami, Florida
  - Winship Cancer Institute at Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Winship Cancer Institute at Emory Saint Joseph's Hospital, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Health Schwarz Cancer Center, Indianapolis, Indiana
  - Indiana University Health - Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Indiana University Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Eastern Maine Medical Center (Northern Light), Brewer, Maine
  - Dana Farber Cancer Institite, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Brigham Cancer Center - Foxborough, Foxborough, Massachusetts
  - Cape Cod Healthcare Center, Hyannis, Massachusetts
  - Dana-Farber at Milford, Milford, Massachusetts
  - Dana-Farber at South Shore Hospital, Weymouth, Massachusetts
  - Dana-Farber Cancer Insitute at Londonderry Hospital, Londonderry, New Hampshire
  - New York University Langone Hospital -Brooklyn, Brooklyn, New York
  - New York University Langone Hospital - Long Island, Mineola, New York
  - New York University Langone Health, New York, New York
  - UNC Rex Hematology Oncology Associated - Cary, Cary, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - UNC Rex Hematology Oncology Associates of Garner, Garner, North Carolina
  - UNC Rex Cancer Center, Raleigh, North Carolina
  - UNC Rex Cancer Center at Wakefield, Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Greco-Hainsworth Centers for Research/Tennessee Oncology, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine Medical Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Waks AG, Chen EL, Graham N, Frey AM, Almeida K, Attaya V, Ryding C, Abbass I, Fung A, Sussell J, Cortazar P, Harvey C, Leth D, Faggen M, Sinclair N, Walsh J, Tung N, Sinclair S, Lo S, Yardley D, Valero V, Meisel J, Ballinger TJ, Adams S, Carey LA, Rauch JK, Abramson VG, Williams NO, Chen WY, Leone JP, Schumer ST, Tayob N, Tolaney SM. Subcutaneous vs Intravenous Trastuzumab/Pertuzumab: A Time and Motion Substudy of a Phase II Trial of Adjuvant Trastuzumab/Pertuzumab for Stage I HER2+ Breast Cancer (ADEPT trial). JCO Oncol Pract. 2025 Mar;21(3):351-357. doi: 10.1200/OP.24.00021. Epub 2024 Jul 19. PMID 39028923